CLINICAL TRIAL: NCT03731520
Title: Determination of Exercise Behavior in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saime Nilay Arman (Other)
Responsible Party: Sponsor-Investigator, Saime Nilay Arman, Assist.Prof., Istanbul University
Organization: Istanbul University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC2
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; exercise; behavior
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing exercise behavior (Experimental): determining exercise behaviour in patients with JIA by using specific scales
  Interventions: Diagnostic Test: Assessing exercise behavior

INTERVENTIONS:
Diagnostic Test: Assessing exercise behavior — 11-point Numeric Analogue Scale (NRS) for satisfaction of exercising, Exercise Stages of Change Scale-Short Form (ESCS), Exercise Self-Efficacy Scale (ESES), and Decisional Balance Scale (DBS) for exercise behaviour will be inquired for the patients with JIA.

SUMMARY:
Juvenile idiopathic arthritis (JIA) is one of the most common rheumatic diseases in childhood, affecting at least 1 in 1000 children. Children with JIA experience joint inflammation and swelling, pain and tenderness, morning stiffness, limited mobility. Children with JIA complain pain and have lower functional ability and decreased quality of life compared with their peers. Many studies have reported that patients with JIA have low physical activity levels and also exercise therapy is considered an important component of the treatment of JIA. Nowadays, studies for evaluating exercise behaviours in order to cope with physical inactivity for many chronic diseases are becoming increasingly important.The objective of this study is to determine exercise behaviour in patients with JIA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as JIA according to ILAR classification
* Aged between 6-18
* Adequate cognitive function for understanding questions

Exclusion Criteria:

- a parent who does not have a smartphone

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
11-point Numeric Analogue Scale | baseline
Exercise Stages of Change Scale-Short Form | baseline
Exercise Self-Efficacy Scale | baseline
Decisional Balance Scale | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No